CLINICAL TRIAL: NCT04084184
Title: An Open-label, Randomized, Single-dose Crossover Study to Evaluate the Pharmacokinetics, Safety and Tolerability of HGP1602 in Healthy Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety and Tolerability of HGP1602 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-DAPA-101
Record Dates: First submitted 2019-09-09; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): Period 1 : Fasted state + HGP1812, Period 2 : Fasted state + HGP1602
  Interventions: Drug: HGP1812; Drug: HGP1602
- Sequence 2 (Experimental): Period 1 :Fasted state + HGP1602, Period 2 : Fasted state + HGP1812
  Interventions: Drug: HGP1812; Drug: HGP1602

INTERVENTIONS:
Drug: HGP1812 — Dapagliflozin (Forxiga) 10mg
Drug: HGP1602 — Dapagliflozin 10mg

SUMMARY:
An open-label, randomized, single-dose crossover study to evaluate the pharmacokinetics, safety and tolerability of HGP1602 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19~45 years in healthy volunteers
2. BMI is more than 18.5 kg/m^2 , no more than 29.9 kg/m^2
3. Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
2. Subjects who judged ineligible by the investigator

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Cmax of Dapagliflozin | pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation
AUClast of Dapagliflozin | pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation

SECONDARY OUTCOMES:
AUCinf of Dapagliflozin | pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation
Tmax of Dapagliflozin | pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation
t1/2 of Dapagliflozin | pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation
CL/F of Dapagliflozin | pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation
Vd/F of Dapagliflozin | pre-dose(0 hour), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hour
  pharmacokinetic evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No